CLINICAL TRIAL: NCT05846425
Title: Investigating the Effect of Yoga-based Breathing Styles on the Human Brain, With a Focus on Memory
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universität des Saarlandes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MST-Breathing Study
Record Dates: First submitted 2023-04-26; First posted 2023-05-06 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Hypoventilation; Hyperventilation
Keywords: Mnemonic similarity task; Yoga-breathing; Memory enhancement
MeSH Terms: conditions — Hypoventilation; Hyperventilation

STUDY DESIGN:
Intervention Model Description: Nose-breathing group, Mouth-breathing group, Control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nose-breathing (Experimental): Controlled nose-breathing
  Interventions: Other: Nose-breathing training
- Mouth-breathing (Active Comparator): Controlled mouth-breathing
  Interventions: Other: Mouth-breathing training
- Control group (No Intervention): no intervention

INTERVENTIONS:
Other: Nose-breathing training — 13 days of controlled nose-breathing training at a specific frequency with a duration of approximately 15 min a day
  Arms: Nose-breathing
Other: Mouth-breathing training — 13 days of controlled mouth-breathing training at a specific frequency with a duration of approximately 15 min a day
  Arms: Mouth-breathing

SUMMARY:
The goal of this clinical trial is to learn if yoga-based breathing styles could improve memory performance in adult persons without relevant prior experience in yoga, meditation or similar disciplines and without existing health problems which could hinder the implementation of the breathing exercises.

The main questions it aims to answer are:

* Can the memory performance get better ?
* Can the subjective stress level be reduced ?

Participants will complete a memory test while doing a specific nasal and oral breathing.

They will complete a two-week training period after the test with daily nasal or mouth breathing training or no training at all, depending on the group, the are divided into.

Researchers will compare the effect of different breathing styles on memory ability among themselves.

DETAILED DESCRIPTION:
The goal of this clinical trial is to learn about the effect of yoga-based breathing styles on the human brain regarding memory performance in adult persons without relevant prior experience in yoga, meditation or similar disciplines and without existing health problems which could hinder the performance of the breathing exercises.

The main questions it aims to answer are:

* Is there an improve of memory performance through performing the controlled yoga-based breathing styles ?
* Is there a relevant reduction of the subjective stress level through performing the controlled yoga-based breathing styles

Participants will complete a memory test while performing controlled nasal and oral breathing.

They will complete a two-week training period after the test with daily nasal or mouth breathing training or no training at all, depending on the group assignment.

Researchers will compare the nasal breathing group to the mouth breathing and the comparison group to see if the nasal breathing results in a significant improvement of the memory capacity.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to take on the 2-week exercises but no new athletic or meditative activities
* Yoga-naive and without significant prior experience in various meditative or athletic disciplines that ostensibly involve elements of breath control
* Access to a device with internet access
* Signing of the consent form to participate in the study

Exclusion Criteria:

* Known clinically relevant internal or neurological diseases, especially if associated with chronic pathological oxygenation (e.g. COPD, severe bronchial asthma, sleep apnea, but also CKD).
* History of drug or alcohol abuse
* Known psychiatric illnesses that currently require therapy (e.g., pronounced claustrophobia)
* Medication that could falsify the data collected
* Lack of consent to take note of possible incidental findings
* known epileptic seizures, which could be intensified by the visual insertion of the stimuli

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-06-03 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Improvement of learned images | 2 weeks
  Memory improvement by performing the home nasal breathing training. The correctness of the mapping is measured by the percentage correctness of the given answers in the memory test, which takes place promptly after the learning phase and 2 weeks later.

SECONDARY OUTCOMES:
Reduction of subjective stress level | 2 weeks
  The subjective stress level is determined by a subjective stress statement, before and after each learning and retrieval phase, at the first appointment and at the second after 2 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Krick, Dr.rer.med., Principal Investigator — University of Saarland
Locations (1):
- Department of Diagnostic and Interventional Neuroradiology, Saarland University Medical Center, Homburg, Saarland, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zelano C, Jiang H, Zhou G, Arora N, Schuele S, Rosenow J, Gottfried JA. Nasal Respiration Entrains Human Limbic Oscillations and Modulates Cognitive Function. J Neurosci. 2016 Dec 7;36(49):12448-12467. doi: 10.1523/JNEUROSCI.2586-16.2016. PMID 27927961
- [Background] Klippenstein JL, Stark SM, Stark CEL, Bennett IJ. Neural substrates of mnemonic discrimination: A whole-brain fMRI investigation. Brain Behav. 2020 Mar;10(3):e01560. doi: 10.1002/brb3.1560. Epub 2020 Feb 3. PMID 32017430
- [Background] Stark SM, Kirwan CB, Stark CEL. Mnemonic Similarity Task: A Tool for Assessing Hippocampal Integrity. Trends Cogn Sci. 2019 Nov;23(11):938-951. doi: 10.1016/j.tics.2019.08.003. Epub 2019 Oct 6. PMID 31597601